CLINICAL TRIAL: NCT00656448
Title: Randomized Study of Procrit vs no Procrit in Patients With Newly Diagnosed Acute Myelogenous Leukemia (AML) or High-risk Myelodysplastic Syndrome (MDS) Undergoing Frontline Myelosuppressive Induction/Consolidation Chemotherapy
Brief Title: A Randomized Trial of Procrit vs. No Procrit in AML and High Risk MDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-0890
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Leukemia
Keywords: Acute Myelogenous Leukemia; AML; Myelodysplastic Syndrome; MDS; Leukemia; Procrit; Epoetin Alfa; Epogen
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procrit Arm (Experimental): Participants receive Procrit along with blood transfusions. Procrit 40,000 units subcutaneously every week starting within two weeks (before or after) from the start of induction chemotherapy.
  Interventions: Drug: Procrit
- No Procrit: Standard Arm (No Intervention): Participants do not receive Procrit before receiving blood transfusions.

INTERVENTIONS:
Drug: Procrit — 40,000 units sq every week starting within two weeks (before or after) from the start of induction chemotherapy.
  Other Names: Epoetin Alfa; Epogen
  Arms: Procrit Arm

SUMMARY:
The goal of this clinical research study is to find out if Procrit (epoetin alfa) will help decrease the need for blood transfusions in patients who have Acute Myelogenous Leukemia (AML) or High-risk Myelodysplastic Syndrome (MDS) and are receiving chemotherapy. Researchers also want to learn about the remission rates (rates of recovery) in patients with cancer who have received treatment with epoetin alfa. The safety and effectiveness of this therapy will also be studied.

DETAILED DESCRIPTION:
Epoetin alfa is a medication that helps the body make more red blood cells. Researchers want to find out if it will be effective in reducing the need for blood transfusions in patients who have AML or high-risk MDS and are receiving chemotherapy.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 treatment groups. Participants in one group will be given epoetin alfa along with blood transfusions, if the doctor thinks it is necessary. Participants in the other group will not receive epoetin alfa. Instead they will only have blood transfusions, which is the standard of care.

No matter what group you are in, you will receive transfusions if your hemoglobin (an element of red blood cells that carries oxygen) drops below a certain level or if the doctor thinks it is necessary. You will be asked to keep a diary listing the dates of all transfusions you receive.

The study doctor will monitor your hemoglobin levels by checking your standard blood tests done by your treating doctor. If your hemoglobin rises above a certain level, treatment with epoetin alfa may be temporarily stopped until your hemoglobin level decreases.

If you are assigned to receive epoetin alfa, you will receive it once a week by subcutaneous (just under the skin) injection during your regularly scheduled chemotherapy. You will receive treatment with epoetin alfa for up to 12 weeks.

If you experience any intolerable side effects or the disease gets worse, you will be taken off this study.

Participants in both groups will continue to receive chemotherapy during this study as regularly scheduled. During chemotherapy (as part of your standard of care), you will have around 1 tablespoon of blood drawn every 1-2 weeks for routine blood tests.

This is an investigational study. Epoetin alfa is FDA approved and commercially available. Up to 54 patients will take part in this study. All will be enrolled at the University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AML or high-risk MDS (based on International Prognostic Scoring System (IPSS): refractory anemia with excess of blasts (RAEB) or RAEB in transformation [RAEB-t]) receiving frontline induction chemotherapy with any high dose or conventional dose cytarabine-containing regimen or clofarabine-containing regimen at MD Anderson Cancer Center.
* Patients must be enrolled on the study within two weeks of the start of induction chemotherapy.
* Patients with documented iron, vitamin B12, or folate deficiency are eligible, but should receive replacement therapy while on study.
* Understand and voluntarily sign an informed consent form.

Exclusion Criteria:

* Patients with prior treatment with any form of erythropoietin within the previous month.
* Patients with uncontrolled hypertension (> or =140/90), uncontrolled, clinically significant cardiac arrhythmias, or history of pulmonary embolism or thrombosis within the last 5 years.
* New onset (within 3 months prior to randomization) or poorly controlled seizures.
* Patients with known hypersensitivity to the active substance or any of the excipients.
* Pregnant or lactating women.
* Acute Erythroleukemia (M6 French-American-British (FAB) classification)
* Hemoglobin greater than or equal to 10g/dl
* Patients with head and neck cancer receiving radiation therapy when erythropoiesis-stimulating agents (ESAs) were given to maintain hemoglobin levels of more than 12 g/dL.
* Patients with metastatic breast cancer receiving chemotherapy when ESAs were given to maintain hemoglobin levels of more than 12 g/dL.
* Patients with chronic kidney failure when ESAs were given to maintain hemoglobin levels of more than 12 g/dL.
* Patients requiring major surgery would be taken off study due to a higher chance of blood clots being reported while taking ESAs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, M.D., Study Chair — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center's Official Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 27, 2008 to February 18, 2010. All recruitment done at the University of Texas (UT) MD Anderson Center.
Pre-assignment Details: Of the 51 participants enrolled for the epoetin alfa (Procrit) study, fifty (50) participants were randomized and one excluded as a screening failure.
Period: Overall Study
Arm/Group | Procrit Arm | No Procrit: Standard Arm
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Procruit: Standard Arm: Participants do not receive Procrit before receiving blood transfusions.
- Total: Total of all reporting groups
Arm/Group | Procrit Arm | No Procruit: Standard Arm | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 61 [22 to 67] | 62 [34 to 79] | 62 [22 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Participant Transfusions Required During 12 Weeks of Treatment
Description: The number and frequency of packed red blood cells (PRBC) transfusions assessed and compared between two groups, treatment group ("Procrit") and standard care group ("No Procrit"). Participants log all PRBC transfusions. Reported are the number of transfusions in the treatment arm during induction and consolidation chemotherapy with the concomitant use of epoetin alfa during therapy, and in the standard arm those that occured during same 12 week period.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: Transfusions per Participant
Arm/Group | Procrit Arm | No Procrit: Standard Arm
Number analyzed (Participants) | 25 | 25
Transfusions per Participant | 7 [1 to 16] | 7 [2 to 13]

2. Secondary Outcome: Number of Participants With Complete Remission
Description: International Working Group (IWG) criteria for responses defined as: Complete Remission (CR) - Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x 10^9/L and platelet count > 100 x 10^9/L, and normal bone marrow differential (< 5% blasts); Partial remission (PR): as CR except for presence of 5-25% marrow blasts and with a decrease of marrow blast at least 50%.
Time Frame: After 1 course of therapy, one course is 4 weeks.
Measure: Number; unit: participants
Arm/Group | Procrit Arm | No Procruit: Standard Arm
Number analyzed (Participants) | 25 | 25
participants
  Complete Remission | 24 | 18
  Early Death | 0 | 3
  Partial Response | 1 | 4

ADVERSE EVENTS:
Time Frame: Participants followed for one month after removal from study following 12 week treatment period. The overall study period was 5 years and 3 months.
Arm/Group | Procrit Arm | No Procruit: Standard Arm
Serious Adverse Events (participants affected / at risk) | 2/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procrit Arm (N=25) | No Procruit: Standard Arm (N=25)
Posterior reversible encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes